CLINICAL TRIAL: NCT04042207
Title: In Adults With Very Unstable Type 1 Diabetes, is the DBLHU Closed-Loop Insulin Delivery System Able to Improve Blood Glycemic Control Compared to Low-Glucose-Predictive-Suspend System: Two-center, Randomized, Open-label Study
Brief Title: Diabeloop for Highly Unstable Type 1 Diabetes
Acronym: DBLHU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019-A01365-52
Record Dates: First submitted 2019-07-19; First posted 2019-08-01 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Brittle; Closed-Loop
Keywords: Artificial pancreas; Very Unstable Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: N-of-1 trials consists in a prospectively planned, multiple crossover study in a single individual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference treatment (Open-Loop) (Active Comparator): Sensor-augmented pump therapy (SAP) namely the Low Glucose Predictive Suspend system or LGPS and a blinded glucose sensor (Dexcom G6) followed by a 48-week extension period in closed-loop condition
  Interventions: Device: Low Glucose Predictive Suspend system; Device: DBLHU System
- DBLHU system (Closed-Loop) (Experimental): DBLHU software (a Model Predictive Control [MPC]-based glucose control algorithm) running on handset associated with the six-generation glucose sensor (Dexcom G6) and Kaleido insulin pump followed by a 48-week extension period in closed-loop condition
  Interventions: Device: DBLHU System

INTERVENTIONS:
Device: Low Glucose Predictive Suspend system — consists of sensor-augmented pump therapy (SAP) / Low Glucose Predictive Suspend system (with predictive low glucose management technology)
  Other Names: Open-loop condition
  Arms: Reference treatment (Open-Loop)
Device: DBLHU System — DBLHU system embeds a regulation algorithm to automatically regulate the patient's glycaemia. It takes as input glycaemia value received every 5 minutes from the CGM and patient inputs related to meals and physical activities and it calculates the amount of insulin to be delivered. It sends this information to the pump that automatically delivers this quantity.
  Other Names: Closed-loop condition

SUMMARY:
Feasibility study, comparing experimental treatment (DBLHU closed-loop system) with reference treatment (Low Glucose Predictive Suspend system) in 7 patients going through a series of N-of-1 trials. Each N-of-1 trial consists in a prospectively planned, multiple crossover study in a single individual. Two blocks of two periods of four weeks each (closed loop or open loop) will be conducted. Within each block, the sequence closed loop-open loop or open loop-close loop is randomized. Outcomes will be analyzed on the third and fourth weeks of period.

A remote monitoring system managed by specialized nurse on behalf of diabetologist, is provided in closed-loop session.

An extension period of 48 weeks with the DBLHU System (closed-loop condition) will be performed at the end of the crossover study phase in real life conditions (without remote monitoring).

ELIGIBILITY:
Inclusion Criteria:

* Subject (aged 22 or more) with Type 1 diabetes for at least 5 years and confirmed C peptide negative
* Treated with continuous subcutaneous insulin infusion (CSII) for ≥ 6 months,
* Trained to carbohydrate counting/flexible insulin therapy,
* Subject that had experienced, despite optimal diabetes management and prior to any equipment with Smartguard technology, glucose instability as defined by at least 2 of the following criteria which would have led to eligibility for pancreatic islet transplantation:

  * occurrence of at least 1 severe hypoglycemic episode during the past 12 months (need for third party),
  * occurrence of ketoacidosis (hospitalization in ICU) without explanation
  * Impaired awareness of hypoglycemia (Clark Score ≥ 4; Gold Score > 4)
  * glucose levels: standard deviation > 50% of the arithmetic mean value on glucose meter or > 40 mg/dl on CGM on a 14-day recording
  * glucose levels: MAGE (mean amplitude of glucose excursions) index > 60 mg/dl
  * glucose levels: coefficient of variation (CV) > 36%
* with persisting extreme glucose variability despite optimal medical care
* with contra-indication or no agreement to undertake pancreatic islet transplantation or pancreas transplantation.
* Subject willing to wear the DBLHU system continuously throughout the study

Exclusion Criteria:

* patient with type 2 diabetes
* age < 22 years old
* patient without any social or familial support able to intervene in case of severe hypoglycemic event
* any permanent and severe condition able to interact with the normal course of the study
* patient with insulin-resistance defined by insulin requirements > 1.5U/kg/d
* patient with a daily dose of insulin required greater than 90 units
* patient receiving a total daily dose of insulin less than 8 U
* use of any insulin that is not 100 U/mL fast-acting insulin analog
* patient suffering from a serious illness or a treatment that might significantly impair diabetes physiology, i.e. glucose-insulin interactions, that might interfere with the medical device (for example irregular treatment of steroids)
* patient having severe problems of uncorrected hearing and/or visual acuity
* patient who is unable to understand and perform all the instructions provided by Diabeloop SA
* patient not willing to perform ≥4 finger stick blood glucose measurements daily
* patients that have frequent exposure to magnetic resonance imaging (MRI), computed tomography (CT) scan, or high-frequency electrical heat (diathermy) treatment.
* patient who has had a pancreatectomy or who has pancreatic malfunctions
* patient having severely altered renal function (Creatinine clearance < 30ml/min)
* patient on dialysis
* pregnancy or breast-feeding patient, or project of pregnancy during the next 6 months
* lack of effective contraception in women of childbearing potential
* all conditions excluding participation to clinical research as defined in France

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Percentage of CGM time in glucose range 70-180 mg/dl, during 24 hours periods for the third and fourth week for each treatment period | 14 days for each treatment period
  Measured by continuous glucose monitoring

SECONDARY OUTCOMES:
Evolution over time of the DBLHU system's performance on a day-to-day and determination of the optimization delay of glycemic control | Over twenty-four hour periods on the four weeks of each treatment period and of the 24-week and 48-week extented CL period.
  Measured by continuous glucose monitoring
Percent of CGM time in glucose range 70-180 mg/dl during nighttime. | Overnight (defined as 00:00 to 06:00) periods on the third and fourth week of each treatment period and during the last 4 weeks of the 24-week and 48-week extented CL period.
  Measured by continuous glucose monitoring
Percent of CGM time in glucose range 70-180 mg/dl during daytime. | Over daytime (defined as 06:00 to 00:00) periods on the third and fourth week of each treatment period and during the last 4 weeks of the 24-week and 48-week extented CL period.
  Measured by continuous glucose monitoring
Percent of CGM time with glucose < 70mg/dl, < 60mg/dl, < 54mg/dl and < 50mg/dl | Over twenty-four hour periods on the third and fourth weeks of each treatment period and during the last 4 weeks of the 24-week and 48-week extented CL period.
  Measured by continuous glucose monitoring
Percent of CGM time with glucose > 180mg/dl, > 250mg/dl, > 300mg/dl and > 360mg/dl | Over twenty-four hour periods on the third and fourth weeks of each treatment period and during the last 4 weeks of the 24-week and 48-week extented CL period.
  Measured by continuous glucose monitoring
Average glycemia level | Over twenty-four hour periods on the third and fourth weeks of each treatment period and during the last 4 weeks of the 24-week and 48-week extented CL period.
  Measured by continuous glucose monitoring
Estimated HbA1c (eHbA1c) levels / glucose management indicator (GMI) | Over twenty-four hour periods on the third and fourth weeks of each treatment period and during the last 4 weeks of the 24-week and 48-week extented CL period.
  Measured by continuous glucose monitoring
HbA1c levels | HbA1c value at the week 24 and week 48 of extented CL period.
  Measured by blood sampling
Glucose coefficient of variation (CV) and Standard deviation (SD) | Over twenty-four hour periods on the third and fourth weeks of each treatment period and during the last 4 weeks of the 24-week and 48-week extented CL period.
  Measured by continuous glucose monitoring
Rate of CGM excursions below 54 mg/dl (3.0 mM) for at least 15 min | Over twenty-four hour periods on the third and fourth weeks of each treatment period and during the last 4 weeks of the 24-week and 48-week extented CL period.
  Mean time spent in hypoglycaemia, defined as sensor glucose values of 54 mg/dL (3∙0 mmol/L) or lower for more than 15 min consecutively
Comparison of MAGE index and Low Blood Glucose Index (LBGI) | Over twenty-four hour periods on the third and fourth weeks of each treatment period and during 24-week extension period
  Mean amplitude of glucose excursions and Low Glucose index as measured by continuous glucose monitoring
Number of acute metabolic events (severe hypoglycemia, severe Diabetic Ketoacidosis [DKA]) | During 4 weeks of each treatment period and during 24-week and 48-week extension period
  Measured by continuous glucose monitoring. Number of severe hypoglycemia is defined as any event requiring third party assistance.
  DKA events. Subjects will be asked to measure blood ketone levels on if their interstitial glucose is above 300 mg/l beyond the usual timeframe following a meal, as part of the safety evaluation for hyperglycemia.
Number of severe hypoglycemia with loss of consciousness | During 4 weeks of each treatment period and during 24-week and 48-week extension period
  Number of severe hypoglycemia with loss of consciousness
Number of hospitalizations for severe hypoglycemia or ketoacidosis | During 4 weeks of each treatment period and during 24-week and 48-week extension period
  Number of hospitalizations
For the use and the acceptance, a satisfaction survey will be done on the daily management of diabetes, the modification of daily life with the system dan the fear of hypoglycemia | after baseline period (2-week); after crossover period; after 24-week and after 48-week extension period
  DTSQ satisfaction questionnaire, with scale from 6 to 0 where 0 is the worth and 6 the best outcome.
Percentage of CGM time in glucose range 70-180 mg/dl, during 24 hours periods | 24-week and 48-week extension period
  Measured by continuous glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Yves BENHAMOU, Pr, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - Grenoble Alpes University Hospital, Grenoble
  - Lille University Hospital, Lille

IPD SHARING:
Plan to Share IPD: No